CLINICAL TRIAL: NCT02823275
Title: Post Operative Evaluation of Quality of Life and Pain in Ankle Fractures: Cast Immobilisation Versus Functional Treatment
Brief Title: Post Operative Quality of Life and Pain in Ankle Fractures: Cast Versus Functional Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator changed jobs
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683-250210-Nicolaas
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Functional mobilisation (Active Comparator)
  Interventions: Other: Functional mobilisation
- plaster cast fixation (Experimental)
  Interventions: Other: Short term plaster cast fixation

INTERVENTIONS:
Other: Functional mobilisation — functional mobilisation
  Arms: Functional mobilisation
Other: Short term plaster cast fixation — 2 weeks cast immobilisation
  Arms: plaster cast fixation

SUMMARY:
Rationale: Ankle fractures are common traumatic lesions. In order to restore the anatomical situation of the ankle joint to prevent posttraumatic arthritis, these fractures often need surgical treatment. Both cast immobilisation and functional treatment have proved to be reliable postoperative treatment regimes. Insight into the quality of life and the level of pain is necessary to determine if these treatments can be related to higher patient satisfaction and earlier resumption of daily activities and work.

Objective: The aim of this study is to examine two postoperative treatments for surgically corrected ankle fractures. Postoperative, direct functional mobilisation is compared to short term plaster cast fixation. The focus of this study is on quality of life, pain and the use of pain medication, and resumption of work and daily activities.

Main study parameters/endpoints:

Quality of life, Function, pain, swelling, daily activities and work, disabilities (pain disability index), complications

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 at the time of surgery
* Ankle fractures needing operative correction
* Weber type B or C, Lauge Hansen type supination-adduction, supination-external rotation and pronation-external rotation
* Closed fractures
* Postoperative stable for exercise
* Operated at the University Medical Centre St Radboud, Nijmegen or Alysis Zorggroep, Rijnstate Hospital, Arnhem

Exclusion Criteria:

* Open fractures
* Fractures with complete dislocation of the ankle joint
* Body Mass Index > 30
* Previous ankle fracture on the affected side
* Concomitant traumatic injuries reducing the ability for postoperative mobilization
* Pre-existent use of pain medication, medication affecting fracture- and wound healing
* Postoperative unstable for exercise
* Co-morbidity: pain syndromes, Fontaine IIB, III and IV, symptomatic venous insufficiency, auto-immune disorders, rheumatic arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
pain | 6 weeks
  Visual Analog Pain Scale
Pain medication used | 6 weeks
  amount of pain medication used

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate, Arnhem, Gelderland
  - Radboud University, Nijmegen, Gelderland